CLINICAL TRIAL: NCT02548091
Title: Evaluation of the Effectiveness of Non-invasive Ventilation on the Reperfusion Pulmonary Oedema Post Pulmonary Artery Angioplasty in the Post Embolic Pulmonary Hypertension
Brief Title: Evaluation of the Effectiveness of Non-invasive Ventilation on the Reperfusion Pulmonary Edema Post Pulmonary Artery Angioplasty in the Post Embolic Pulmonary Hypertension
Acronym: OPR_VNI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-A00399-40
Record Dates: First submitted 2015-09-03; First posted 2015-09-14 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-02

CONDITIONS: Reperfusion Pulmonary Edema
Keywords: non invasive ventilation; reperfusion pulmonary edema; chronic thrombolic pulmonary hypertension; pulmonary artery angioplasty
MeSH Terms: interventions — Blood Specimen Collection; Interleukin-8; Interleukin-10; Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preventive non invasive ventilation (Active Comparator): Patients will receive the non invasive ventilation (NIV) systematically during the whole procedure of pulmonary angioplasty, and then systematically in post procedure period, 1 hour every 4 hours, during the whole hospitalization in post anesthesia care unit (PACU).
  Interventions: Other: Blood samples for assays of plasma inflammatory markers (cytokines InterLeukin-6, InterLeukin-8, InterLeukin-10); Procedure: Non invasive ventilation; Procedure: monitoring system Pulse-Induced Contour Cardiac Output (Picco); Procedure: Computed tomography (CT)
- Non invasive ventilation on demand (Other): Patients will not receive the NIV during the procedure of pulmonary angioplasty; in case of respiratory decompensation in post procedure period they will receive NIV during the whole hospitalization in PACU according to the following criteria: paradoxical breathing, respiratory rate above 25/minutes, a ratio of arterial oxygen pressure to fraction of inspired oxygen values (PaO2/FiO2) below 200.
  Interventions: Other: Blood samples for assays of plasma inflammatory markers (cytokines InterLeukin-6, InterLeukin-8, InterLeukin-10); Procedure: Non invasive ventilation; Procedure: monitoring system Pulse-Induced Contour Cardiac Output (Picco); Procedure: Computed tomography (CT)

INTERVENTIONS:
Other: Blood samples for assays of plasma inflammatory markers (cytokines InterLeukin-6, InterLeukin-8, InterLeukin-10) — The same amount of blood sample is collected from both arms of study at the same time of the procedure.
  In each patient, in the per procedure period, a total of 50 milliliters of blood sample is drawn from the pulmonary circulation downstream and upstream of obstructive lesion, the trunk of pulmonary artery, the superior vena cava and the femoral arterial line prior to angioplasty and at the end of procedure; in the post interventional care unit 10 milliliters of blood sample will be draw daily from the superior vena cava catheter line and femoral arterial line.
Procedure: Non invasive ventilation
Procedure: monitoring system Pulse-Induced Contour Cardiac Output (Picco)
Procedure: Computed tomography (CT)

SUMMARY:
The purpose of this study is to determine whether Non Invasive Ventilation are effective in prevention of reperfusion pulmonary edema after pulmonary artery angioplasty. Our hypothesis is that administration of Non Invasive Ventilation during the procedure and systematically in post procedure period is a protective factor against the development and severity of reperfusion pulmonary edema.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* First and /or second procedure of pulmonary artery angioplasty
* Mean pulmonary arterial pressure ≥ 40 mmHg and/or pulmonary vascular resistance ≥ 8 WU (Wood unit)
* Patient who signed informed consent
* Patients affiliated to a social security program

Exclusion criteria:

* severe neurological disease: Coma Glasgow Scale < 8, severe cognitive decline, postural instability, loss of autonomy.
* psychiatric disease (illness)
* sepsis, severe sepsis and septic shock, according to definitions and diagnostic criteria for sepsis of 'Surviving Sepsis Campaign 2012'
* severe respiratory failure defined by a total lung capacity (TLC)< 50% of the predicted value and/or expiratory volume in 1 second (FEV) < 30% of predicted value
* obstructive sleep apnea syndrome with Continuous Positive Airway treatment
* preexisting hemorrhagic syndrome or coagulation factors deficiency
* severe renal insufficiency with glomerular filtration rate < 30 ml/min
* severe hepatic failure with hepatic encephalopathy, hemodynamic disorder, decompensates cirrhosis, metabolic disorder( metabolic acidosis, hypoglycemia) hepatorenal syndrome, coagulation disorder (factor V< 50%,disseminated intravascular coagulation)
* patient refusal of participation in the study program
* subjects not affiliated to social security program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Lung Injury Score. | Daily during hospitalization in the PACU on day 1 to 7.

SECONDARY OUTCOMES:
Assays of plasma inflammatory markers (InterLeukin-6 , IInterLeukin-8, InterLeukin-10). | 2 years
  The concentration will be given in pg/mL
Extravascular Lung Water (EVLW) measures. | 2 years
  EVLW is measure by thermodilution technique using a Pulse-Induced Contour Cardiac Output system (PICCO). The unit of EVLW is mL/Kg
Computed tomography (CT) score | 2 years
Doppler pulsatility of the portal vein and its pulsatility ratio | 2 years
Pulmonary Vascular Index (PVI) measures | 2 years
  PVI is measure by thermodilution technique using a Pulse-Induced Contour Cardiac Output system (PICCO

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France